CLINICAL TRIAL: NCT06818513
Title: Effects of Gastrostomy and Intermittent Oral Tube Feeding on Patients With Dysphagia After Stroke
Brief Title: Effects of Gastrostomy and Oral Tube Feeding on Patients With Dysphagia After Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, The Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PEG in stroke dysphagia
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Gastrostomy; Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral tube group+routine rehabilitation therapy (Experimental): All patients are provided with routine rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  The oral tube group will be given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups.
  Interventions: Behavioral: routine rehabilitation therapy; Dietary Supplement: Oral tube feeding
- Gastrostomy group+routine rehabilitation therapy (Active Comparator): All patients were provided with routine rehabilitation therapy as follows:
  Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  The Gastrostomy group will be given enteral nutritional support with Gastrostomy. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Behavioral: routine rehabilitation therapy; Dietary Supplement: Gastrostomy

INTERVENTIONS:
Behavioral: routine rehabilitation therapy — Including： Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
Dietary Supplement: Gastrostomy — Feeding begins through the gastrostomy tube. A registered dietitian will develop a tailored feeding plan, specifying the type and amount of nutrition. Healthcare providers regularly monitor the patient's tolerance to feeding, checking for any signs of complications. Adjustments to the feeding regimen may be made based on the patient's progress and nutritional needs.
  Arms: Gastrostomy group+routine rehabilitation therapy
Dietary Supplement: Oral tube feeding — During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Arms: Oral tube group+routine rehabilitation therapy

SUMMARY:
The goal of this clinical trial is to compare the differences in swallowing function, quality of life and nutritional status between ischemic stroke patients with dysphagia using Intermittent Oro-esophageal Tube and Gastrostomy. Patients will be randomly divided into an oral tube group and a Gastrostomy group, all receiving routine rehabilitation treatment. On this basis, the oral tube group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the Gastrostomy group will use Gastrostomy. Researchers will compare changes in swallowing function, quality of life and nutritional status of two groups of patients before and after the study to see if Intermittent Oro-esophageal Tube can improve the quality of life and nutritional status between ischemic stroke patients compared Gastrostomy.

DETAILED DESCRIPTION:
This study will last 15 days for each patient. The goal of this clinical trial is to compare the differences in swallowing function, quality of life and nutritional status between ischemic stroke patients with dysphagia using Intermittent Oro-esophageal Tube and Gastrostomy. Patients will be randomly divided into an oral tube group and a Gastrostomy group, all receiving routine rehabilitation treatment. On this basis, the oral tube group will use Intermittent Oro esophageal Tube for enteral nutrition support, while the Gastrostomy group will use Gastrostomy. Researchers will compare changes in swallowing function, quality of life and nutritional status of two groups of patients before and after the study to see if Intermittent Oro-esophageal Tube can improve the quality of life and nutritional status between ischemic stroke patients compared Gastrostomy.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Meeting the diagnostic criteria for ischemic stroke .
* Dysphagia confirmed by Videofluoroscopic Swallowing Study.
* Clear consciousness.
* No history of prior stroke.
* Stable vital signs.

Exclusion Criteria:

* Use of tracheostomy tubes.
* Dysphagia that might be caused by other diseases that might cause dysphagia, such as head and neck tumors, traumatic brain injury, myasthenia gravis, etc.
* Complicated with severe liver and kidney failure, tumors, or hematological disorders.
* Simultaneously in need to undergo other therapy that might affect the outcomes of this study.
* Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Body mass index | day 1 and day 15
  body mass index will be calculated as body weight/height^2.

SECONDARY OUTCOMES:
Dysphagia Handicap Index | day 1 and day 15
  The Dysphagia Handicap Index is a 25-item scale to evaluate swallowing-related quality of life. The scale scores range between 0 to 100 and a higher score indicate poorer quality of life
Penetration-Aspiration Scale | day 1 and day 15
  The Penetration-Aspiration Scale was used to evaluate airway protection. The score could range between 0 and 8, with higher scores indicating poor swallowing safety.
Modified Barium Swallow Impairment Profile | day 1 and day 15
  The Modified Barium Swallow Impairment Profile was conducted by an independent and registered speech-language pathologist. The scale includes 17 items to cover oral, pharyngeal, and esophageal phases of swallowing. The total score ranges from 0 to 55, with higher scores indicating poorer swallowing function.